CLINICAL TRIAL: NCT05571007
Title: Effect of Acupressure on Fatigue in Hemodialysis Patients: A Single-blinded Randomized Controlled Trial
Brief Title: Effect of Acupressure on Fatigue in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Woung-Ru Tang (Other)
Collaborators: Harapan Bangsa University (Unknown); RS Prof. Dr. Margono Soekardjo Purwokerto (Unknown)
Responsible Party: Sponsor-Investigator, Woung-Ru Tang, Professor, Chang Gung University
Organization: Chang Gung University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3010/KEPK/VII/2019
Record Dates: First submitted 2022-09-30; First posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: End-stage Renal Disease
Keywords: End-stage renal disease; Hemodialysis; Acupressure; Fatigue; Sleep; Anxiety/depression
MeSH Terms: conditions — Kidney Failure, Chronic; Fatigue; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- True acupressure (Experimental): Using three true acupoints. Acupoints: Yongquan (K1), Sayingjiao (SP6), Zusanli (ST36). Patient Position: Lying or sitting position. Time: first 2 hours of HD.
  Interventions: Other: True acupressure
- Sham acupressure (Sham Comparator): Using three sham acupoints. Acupoints: Sham acupoints are located on 1 cun from the true acupoint. Patient Position: Lying or sitting position. Time: first 2 hours of HD.
  Interventions: Other: Sham acupressure

INTERVENTIONS:
Other: True acupressure — Duration: 3 minutes for each acupoint, applied bilaterally (right and left sides).
  Total time: 18 minutes/acupressure therapy.
  Arms: True acupressure
Other: Sham acupressure — Duration: 3 minutes for each acupoint, applied bilaterally (right and left sides).
  Total time: 18 minutes/acupressure therapy.
  Arms: Sham acupressure

SUMMARY:
OBJECTIVE: To investigate the effect of acupressure on fatigue in patients with end-stage renal disease (ESRD) undergoing hemodialysis (HD) as well as assess sleep quality and psychological status HYPOTHESIS TO BE TESTED: Upon intervention completion, the experimental group will exhibit lower severity of fatigue and depression/anxiety and improved sleep quality compared to the control group.

DESIGN AND SUBJECTS: A randomized controlled trial with experimental and control groups. A total of 116 patients with ESRD who screen positive for fatigue severity ≥ 4 (using a single-item indicator of fatigue, which ranges from 0 to 10 points) will be recruited.

STUDY INSTRUMENTS: Brief Fatigue Inventory (BFI), Pittsburgh Sleep Quality Index (PSQI), and Hospital Anxiety and Depression Scale (HADS) INTERVENTION: A 4-week acupressure intervention was performed by the principal investigator (PI) for every subject by applying the rate of two rotations per second, three times a week.

MAIN OUTCOME MEASURES: Primary: fatigue. Secondary: sleep quality, depression, and anxiety.

DATA ANALYSIS: Multiple regression was used to analyze between-group differences in BFI and PSQI, while ordinal logistic regression was used to analyze the subscales of the HADS.

EXPECTED RESULTS: The proposed acupressure intervention is useful for alleviating fatigue and related symptoms (sleep quality, depression, and anxiety) experienced by patients with ESRD.

DETAILED DESCRIPTION:
The prevalence and impact of fatigue and related symptoms in patients with ESRD have been clearly demonstrated in the literature, which also emphasizes the need for evidence-based interventions targeting symptom management in such patients. The main challenge is identifying an intervention that is not only effective in managing hemodialysis-related symptoms, but also feasible, acceptable, and safe for this patient group. The proposed study primarily aims to test the effects of acupressure intervention on fatigue in ESRD patients receiving HD using the robust study design of a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≧ 18 years
* 2. HD therapy for at least 3 months
* 3. Experience of fatigue (fatigue severity ≥ 4, using a single-item indicator of fatigue, ranging from 0 to 10 points)
* 4. Absence of lower limb wounds
* 5. Did not receive any complementary treatment

Exclusion Criteria:

* 1. Diagnosis of major depression or psychiatric disorders
* 2. Wound or amputation of the lower extremities, rheumatoid arthritis, or limb fracture

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Brief Fatigue Inventory (BFI) | Before the intervention (baseline, T0)
  A questionnaire will be used to measure the severity of fatigue in the past 24 hours. This 9-item self-reported questionnaire is scored on a 0-10 numerical rating scale, where 0 and 10 represent absence and the highest severity of fatigue, respectively. The BFI score is classified into mild (1-3 points), moderate (4-6 points), and severe fatigue (7-10 points).
Brief Fatigue Inventory (BFI) | Completion of the 4-week intervention (post-test, T1)
  A questionnaire will be used to measure the severity of fatigue in the past 24 hours. This 9-item self-reported questionnaire is scored on a 0-10 numerical rating scale, where 0 and 10 represent absence and the highest severity of fatigue, respectively. The BFI score is classified into mild (1-3 points), moderate (4-6 points), and severe fatigue (7-10 points).

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | Before the intervention (baseline, T0)
  This 19-item self-reported questionnaire is combined to form seven component scores (subjective sleep quality, latency, duration, habit efficiency, disturbances, medication, and daytime dysfunction). Each of these has a range of 0-3 points added to yield a global score with a range of 0-21. A global score higher than five indicates poor sleep quality.
Pittsburgh Sleep Quality Index (PSQI) | Completion of the 4-week intervention (post-test, T1)
  This 19-item self-reported questionnaire is combined to form seven component scores (subjective sleep quality, latency, duration, habit efficiency, disturbances, medication, and daytime dysfunction). Each of these has a range of 0-3 points added to yield a global score with a range of 0-21. A global score higher than five indicates poor sleep quality.
Hospital Anxiety and Depression Scale | Before the intervention (baseline, T0)
  This 14-item questionnaire will be used to measure psychological status. This 14-item questionnaire has two subscales: anxiety (seven items) and depression (seven items). It is measured on a 4-point Likert scale ranging from 0 (not at all) to 3 (very often), with higher scores indicating an increased level of anxiety/depression. The HADS score is classified as severe (16-21 points), moderate (11-15 points), mild (8-10 points), or no anxiety or depression (≤7 points). It is a valid, trustworthy, and easy measurement tool used by health care providers to identify and quantify anxiety and depression.
Hospital Anxiety and Depression Scale | Completion of the 4-week intervention (post-test, T1)
  This 14-item questionnaire will be used to measure psychological status. This 14-item questionnaire has two subscales: anxiety (seven items) and depression (seven items). It is measured on a 4-point Likert scale ranging from 0 (not at all) to 3 (very often), with higher scores indicating an increased level of anxiety/depression. The HADS score is classified as severe (16-21 points), moderate (11-15 points), mild (8-10 points), or no anxiety or depression (≤7 points). It is a valid, trustworthy, and easy measurement tool used by health care providers to identify and quantify anxiety and depression.

CONTACTS AND LOCATIONS:
Overall Officials: Made Suandika, PhDCandidate, Principal Investigator — School of Nursing, Harapan Bangsa University, Central Java, Indonesia
Locations (1):
- RS Prof Dr Margono Soekardjo Purwokerto, Purwokerto, Central Java, Indonesia

REFERENCES:
- [Derived] Suandika M, Chen SY, Fang JT, Yang SH, Tsai YF, Weng LC, Tsay PK, Tang WR. Effect of Acupressure on Fatigue in Hemodialysis Patients: A Single-Blinded Randomized Controlled Trial. J Integr Complement Med. 2023 Feb;29(2):111-118. doi: 10.1089/jicm.2022.0644. Epub 2022 Nov 22. PMID 36413013